CLINICAL TRIAL: NCT04079712
Title: A Phase 2 Study of XL184 (Cabozantinib) in Combination With Nivolumab and Ipilimumab for the Treatment of Poorly Differentiated Neuroendocrine Carcinomas
Brief Title: Testing the Combination of XL184 (Cabozantinib), Nivolumab, and Ipilimumab for Poorly Differentiated Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-05864; NCI-2019-05864 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10315 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10315 (Other: CTEP); UM1CA186689 (NIH); UM1CA186691 (NIH)
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Large Cell Neuroendocrine Carcinoma; Metastatic Neuroendocrine Carcinoma; Metastatic Neuroendocrine Neoplasm; Metastatic Small Cell Neuroendocrine Carcinoma
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Neuroendocrine Tumors; Small Cell Lung Carcinoma | interventions — cabozantinib; Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (cabozantinib s-malate, nivolumab, ipilimumab) (Experimental): Patients receive cabozantinib s-malate PO QD on days 1-21 of cycles 1-4 and days 1-28 of subsequent cycles, nivolumab IV over 30 minutes on day 1, and ipilimumab IV over 90 minutes on day 1 of cycles 1-4 only. Treatment repeats every 21 for 4 cycles then every 28 days for subsequent cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase II trial studies how well the combination of XL184 (cabozantinib), nivolumab, and ipilimumab work in treating patients with poorly differentiated neuroendocrine tumors (i.e., neuroendocrine tumor that does not look like the normal tissue it arose from). Cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving cabozantinib, nivolumab and ipilimumab may shrink the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the overall response rate (ORR) associated with the combination of XL184 (cabozantinib), nivolumab, and ipilimumab in patients with advanced poorly-differentiated neuroendocrine carcinomas (NECs), after the failure of at least one line of prior therapy.

SECONDARY OBJECTIVES:

I. To evaluate progression-free survival (PFS). II. To measure the safety and tolerability of the combination of XL184 (cabozantinib), nivolumab, and ipilimumab in patients with advanced, poorly-differentiated NECs.

III. To evaluate disease control rate (DCR). IV. To measure duration of response (DOR). V. To describe the tumor molecular profile using whole exome sequencing (WES) and correlate it with treatment outcome.

VI. To describe the tumor molecular profile using ribonucleic acid (RNA) sequencing (RNAseq) and correlate it with treatment outcome.

EXPLORATORY OBJECTIVES:

I. To measure the tumor-infiltrating CD8+ T lymphocytes in pre- and on-treatment biopsies.

II. To measure tumor-infiltrating myeloid derived suppressor cells (MDSCs) in pre- and on-treatment biopsies.

III. To measure tumor-infiltrating tumor-associated macrophages (TAM) in the pre and on-treatment biopsies.

IV. To measure the expression of programmed death-ligand 1 (PD-L1) in tumor cells and infiltrating immune cells.

OUTLINE:

Patients receive cabozantinib s-malate orally (PO) once daily (QD) on days 1-21 of cycles 1-4 and days 1-28 of subsequent cycles, nivolumab intravenously (IV) over 30 minutes on day 1, and ipilimumab IV over 90 minutes on day 1 of cycles 1-4 only. Treatment repeats every 21 for 4 cycles then every 28 days for subsequent cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic, histologically confirmed poorly-differentiated neuroendocrine neoplasms per 2018 World Health Organization (WHO) classification, with the exception of small cell lung cancer and merkel cell carcinoma. All variations of poorly differentiated neuroendocrine carcinoma (small cell, large cell and mixed cells) are eligible
* Failure of only one line of prior systemic cancer treatment
* Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
* Patients must have lesions that can be safely biopsied and be willing to have a pre-treatment and an on-treatment biopsy (after 1 month of treatment with the combination regimen) and a blood collection at baseline
* Prior systemic cancer therapy must have been completed at least 4 weeks prior to cycle 1 day 1 of treatment with the combination regimen
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL without granulocyte-colony stimulating (GCSF) factor support
* Hemoglobin >= 9 g/dL
* Serum thyroid stimulating hormone (TSH) within institutional normal limits
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN); =< 3.0 x ULN for patients with Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional ULN
* Alkaline phosphatase =< 3.0 x institutional ULN; =< 5.0 x ULN with documented bone metastases
* Creatinine =< institutional ULN OR creatinine clearance (CrCl) >= 50 mL/min/1.73 m^2 (using the Cockcroft-Gault formula)
* Serum albumin >= 2.8 g/dL
* Lipase < 2.0 x ULN and no radiologic or clinical evidence of pancreatitis
* Urine protein/creatinine ratio (UPCR) =< 1 mg protein/mg creatinine
* Serum phosphorus, calcium, magnesium, and potassium within institutional normal limits
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) test < 1.3 x ULN
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy utilizing agents that do not strongly induce or inhibit cytochrome P450 (CYP) 3A4 with undetectable viral load within 6 months prior to study registration are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression and are off steroid support for at least 4 weeks after treatment for metastases is complete and within 28 days prior to the first dose of study treatment. Radiotherapy should have been stopped at least 4 weeks prior to study registration. Brain surgery should not have occurred within 3 months of study registration to be eligible
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* The effects of XL184 (cabozantinib), nivolumab, and ipilimumab on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. WOCBP should use an adequate method to avoid pregnancy for 5 months after the last dose of study therapy. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity: 25 IU/L or equivalent units of human chorionic gonadotropin [hCG]) within 24 hours prior to the start of study therapy. Women must not be breastfeeding. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of < 1% per year. Men who receive study therapy and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of study therapy. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level < 40 mIU/mL. WOCBP and men who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 5 and 7 months, respectively, after the last dose of study therapy. These durations have been calculated using the upper limit of the half-life for nivolumab (25 days) and are based on the protocol requirement that WOCBP use contraception for 5 half-lives plus 30 days and men who are sexually active with WOCBP use contraception for 5 half-lives plus 90 days. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she (or the participating partner) must inform the treating physician immediately
* Patients must be able to swallow tablets
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients must not require systemic corticosteroids treatment (>= 10 mg/day prednisone equivalents) or other immunosuppressive medications within 28 days prior to study drug administration. Inhaled or topical steroids and adrenal replacement doses < 10 mg/day prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids in patients with adrenal insufficiency are permitted, even if >= 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted, as is steroid pre-medication for contrast allergy
* Patients must not have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T cell co-stimulation or immune checkpoint pathways
* Patients must not have had prior treatment with XL184 (cabozantinib), or any MET-targeting tyrosine kinase inhibitor (TKI), or any MET-targeting monoclonal antibody (MetMAb), such as onartuzumab
* Patients must not have received radiation therapy to any part of the body within 28 days
* Patients must not have clinically relevant, ongoing complications from prior radiation therapy. No radiation therapy is allowed while the patient is on study. Palliative radiation therapy, if needed, should be completed at least 28 days prior to enrollment into the study as described above
* Patients must not require concomitant treatment with oral anticoagulants (e.g., warfarin, direct thrombin, and factor Xa inhibitors) or platelet inhibitors (e.g., clopidogrel). The following anticoagulants are allowed:

  * Low-dose aspirin for cardioprotection (per local applicable guidelines),
  * Low-dose low molecular weight heparins (LMWH),
  * Therapeutic doses of LMWH are allowed in patients without known brain metastases who are on a stable dose of LMWH for at least 6 weeks before the first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor
* Patients must not have had major surgery (e.g., gastrointestinal [GI] surgery or removal or biopsy of brain metastasis) within 4 weeks before first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before the first dose of study treatment and from minor surgery (e.g., simple excision or tooth extraction) at least 10 days before the first dose. Patients with clinically relevant ongoing complications from prior surgery are not eligible
* Patients must not have received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies) within 4 weeks, or nitrosoureas/ mitomycin C within 4 weeks, before the first dose of study treatment. Patients may continue on bone-modifying agents (denosumab or bisphosphonates) with caution
* Patients who have not recovered to baseline from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) according to Common Terminology Criteria for Adverse Events (CTCAE) version (v)0.5 unless the adverse events (AEs) are clinically nonsignificant and/or stable on supportive therapy, with the exception of alopecia
* Patients who are receiving any other investigational agents. Patients must not have received any other type of investigational agent within 4 weeks before the first dose of study treatment to be eligible
* Patients must not have a corrected QT interval calculated by the Fridericia formula (QTcF) > 500 msec by electrocardiogram (EKG) within 28 days before the first dose of study treatment

  * Note: If a single EKG shows a QTcF with an absolute value > 500 msec, two additional EKGs at intervals of approximately 3 min must be performed within 30 min after the initial EKG, and the average of these three consecutive results for QTcF will be used to determine eligibility
* Patients should not have known, untreated brain metastases or leptomeningeal metastases because of poor prognosis and concerns that progressive neurologic dysfunction could confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study
* Patients must not have a history of severe hypersensitivity reactions to any monoclonal antibodies
* Patients must not require concomitant treatment with strong CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, or St. John's wort). Because lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, patients will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients must not have uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association (NYHA) Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment within seven days prior to the first dose of study treatment.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis [DVT], pulmonary embolism [PE]) within 6 months before first dose.
  * GI disorders including those associated with a high risk of perforation or fistula formation:

    * The patient has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
    * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. Complete healing of an intra-abdominal abscess must be confirmed before first dose.
  * Clinically significant hematuria, hematemesis, or hemoptysis or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose.
  * Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
  * Lesions invading or encasing any major blood vessels.
  * Other clinically significant disorders that would preclude safe study participation.

    * Serious non-healing wound/ulcer/bone fracture.
    * Uncompensated/symptomatic hypothyroidism.
    * Moderate to severe hepatic impairment (Child-Pugh B or C).
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because XL184 (cabozantinib) has the potential for teratogenic or abortifacient effects, and the effects of nivolumab and ipilimumab on the developing fetus are not well known. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother, breastfeeding must be discontinued if the mother is treated with XL184 (cabozantinib), nivolumab, or ipilimumab
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including high dose systemic corticosteroids, should be excluded. These include but are not limited to: immune-related neurologic disease, such as multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, or myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, or autoimmune hepatitis. Patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patients with vitiligo, type I diabetes mellitus (DM), or endocrine deficiencies (e.g., thyroiditis) managed with replacement hormones, including physiologic corticosteroids, are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication, and patients with positive serology, (e.g., antinuclear antibodies [ANA] or anti-thyroid antibodies) should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2026-08-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anteneh A Tesfaye, Principal Investigator — Yale University Cancer Center LAO
Locations (46):
- United States (45):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Farmington Health Center, Farmington, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab): Patients receive cabozantinib s-malate PO QD on days 1-21 of cycles 1-4 and days 1-28 of subsequent cycles, nivolumab IV over 30 minutes on day 1 all cycles, and ipilimumab IV over 90 minutes on day 1 of cycles 1-4 only. Treatment repeats every 21 days for 4 cycles then every 28 days for subsequent cycles in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Started | 17
Completed | 16
Not Completed | 1
Not completed — Disease progression before starting treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: Years] | 62 [27 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17
Weight [Median (Full Range); unit: kilogram (kg)] | 88 [37.1 to 119.5]
Body Surface Area (BSA) [Median (Full Range); unit: meters squared (m^2)] | 2.0 [1.4 to 2.5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: Participants who are considered to have a response are those with either a complete response (CR) (disappearance of all target lesions) or a partial response (PR) (>=30% decrease in the sum of the longest diameter of target lesions) using Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 and assessed by CT or MRI scan.
Time Frame: Up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 16
Participants
  Response | 2
  No Response | 14

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression is defined as a >= 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) and assessed by CT or MRI scan. The duration is from the date of registration to the time of progression or death, whichever occurs first.
Time Frame: Up to 3.5 years
Measure: Median (Full Range); unit: Days
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 16
Days | 85 [23 to 902]

3. Secondary Outcome: Number of Participants Reporting Adverse Events
Description: Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) 5.0 criteria. The population is defined as all patients who have received the study treatment. The highest grade is reported.
Time Frame: Up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 16
Participants
  Grade 5 | 0
  Grade 4 | 3
  Grade 3 | 7
  Grades 1-2 | 6

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR will be defined as the achievement of Complete Response (CR) (disappearance of all target lesions), Partial Response (PR) (>=30% decrease in the sum of the longest diameter of target lesions), or Stable Disease (SD) (between < 30% decrease and >20% increase in the sum of the longest diameter of target lesions) using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT or MRI scan.
Time Frame: Up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 16
Participants
  Achieved disease control | 9
  Did not achieve disease control | 7

5. Secondary Outcome: Duration of Response (DOR)
Description: The time when measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented.
Time Frame: Up to 3.5 years
Measure: Median (Full Range); unit: Days
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 2
Days | 664 [504 to 824]

6. Other Pre Specified Outcome: CD8+ T Lymphocytes
Description: Expression of CD8+ T lymphocytes in the tumor tissue at baseline and during treatment.
Time Frame: Up to Day 35
Population: This biomarker assay was not performed as there were insufficient samples available to interpret the planned correlative studies.
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Myeloid-Derived Suppressor Cells
Description: Presence of myeloid derived suppressor cells in the tumor before and during treatment.
Time Frame: Up to Day 35
Population: as for outcome 6
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Tumor-associated Macrophages
Description: Presence of tumor-associated macrophages in the tumor at baseline and during treatment.
Time Frame: Up to Day 35
Population: as for outcome 6
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: About 3.5 years
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
All-Cause Mortality (participants affected / at risk) | 13/17
Serious Adverse Events (participants affected / at risk) | 10/17
Other Adverse Events (participants affected / at risk) | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab) (N=17)
Pericardial effusion (Cardiac disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 2
Appendicitis (Infections and infestations) | 1
Cholangitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Stoma site infection (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab) (N=17)
Anemia (Blood and lymphatic system disorders) | 6
Sinus bradycardia (Cardiac disorders) | 3
Sinus tachycardia (Cardiac disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 5
Dry eye (Eye disorders) | 1
Vision Changes (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Anal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 7
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 2
Rectal hemorrhage (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Chills (General disorders) | 3
Edema limbs (General disorders) | 5
Fatigue (General disorders) | 10
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 2
Jaw pain (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 3
Covid-19 (Infections and infestations) | 1
Gum infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 11
Alkaline phosphatase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 10
Blood bilirubin increased (Investigations) | 4
Blood lactate dehydrogenase increased (Investigations) | 2
Creatinine increased (Investigations) | 4
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Fibrinogen decreased (Investigations) | 1
GGT increased (Investigations) | 2
Hemoglobin increased (Investigations) | 1
INR increased (Investigations) | 1
Lipase increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 7
Serum amylase increased (Investigations) | 2
Thyroid stimulating hormone increased (Investigations) | 2
Weight loss (Investigations) | 6
White blood cell decreased (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Muscle cramp (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 4
Hypersomnia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Dysuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Hair color change (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Nail changes (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT04079712/Prot_SAP_001.pdf
  • Informed Consent Form (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT04079712/ICF_002.pdf